CLINICAL TRIAL: NCT04560140
Title: Promoting Community Reintegration Using Narratives and Skills Building for Young Adults With Stroke
Brief Title: Promoting Community Reintegration for Young Adults With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Suzanne HS Lo, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NSI
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Stroke; Community reintegration; Narrative; Skill building
MeSH Terms: conditions — Stroke; Narration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Eligible participants will be randomly assigned to receive usual care with the novel 24-week Narrative and Skills-building Intervention.
  Interventions: Behavioral: Narrative and Skills-building Intervention
- Usual care group (No Intervention): Participants will receive usual stroke care.

INTERVENTIONS:
Behavioral: Narrative and Skills-building Intervention — The intervention is grounded in Narrative Theory and Bandura's principles of Self-efficacy and Outcome Expectation. It will consist of eight individual sessions over six months delivered by a facilitator. Participants will be facilitated to narrate their survival experiences and rebuild core life skills.
  Arms: Intervention group

SUMMARY:
This project will investigate the effects of a Narrative and Skills-building Intervention on young stroke survivors' community reintegration and psychosocial outcomes. A randomised controlled trial will be conducted. This is a novel trial to test the short and long-term effects of a theory-based intervention on young stroke survivors' community reintegration.

DETAILED DESCRIPTION:
This project will investigate the effects of a Narrative and Skills-building Intervention on young stroke survivors' community reintegration and psychosocial outcomes. A randomised controlled trial will be conducted. Participants will be facilitated to narrate their survival experiences and rebuild core life skills. Outcomes including community reintegration, depressive symptoms, health-related quality of life, self-efficacy, outcome expectation and satisfaction with performance of self-management behaviours will be measured. This is a novel trial to test the short and long-term effects of a theory-based intervention on young stroke survivors' community reintegration.

ELIGIBILITY:
Inclusion Criteria:

* (1) are 18-64 years of age,
* (2) have a clinical diagnosis of first-ever or recurrent ischaemic or haemorrhagic stroke,
* (3) are living at home after discharge from hospital,
* (4) have a Montreal Cognitive Assessment score >20,
* (5) have a modified Rankin Scale score ≥3,
* (6) can communicate in Cantonese, and
* (7) are able to attend all intervention sessions.

Exclusion Criteria:

* 1) transient ischaemic attack, subdural or epidural haemorrhage,
* 2) experienced cerebrovascular events due to tumours or head trauma,
* 3) mental condition such as depression, schizophrenia, bipolar or personality disorder,
* 4) incomprehensible speech or difficulty in comprehending conversations, or
* 5) have received a self-management programme in the past.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the participants' level of community reintegration | Change from baseline (T0) to immediately (T1), 6 months (T2) and 12 months (T3) after completion of the intervention
  The Chinese version of the Reintegration to Normal Living Index (RNIL-C) will be used to assess the participants' level of community reintegration. It consists of 11 items in eight domains: mobility, self-care, daily work and school activity, recreational and social activities, family roles, personal relationships, presentation of self to others and general coping skills. Participants are asked to rate the extent to which each item describes their situation on a scale from 1 - 'a small extent' to 5 - 'a great extent'. The total score is calculated by summation and normalised to give 100 with a total score range of 25 to 100. A higher score indicates better community reintegration. The RNIL-C has high internal consistency (Cronbach's alpha=0.92) and good convergent validity.

SECONDARY OUTCOMES:
Change in the participants' level of depressive symptoms | Change from baseline (T0) to immediately (T1), 6 months (T2) and 12 months (T3) after completion of the intervention
  The Chinese version of the 15-item Geriatric Depression Scale (GDS) will be used to measure participants' depressive symptoms. Studies support its utility in younger adults (>18 years old), with good diagnostic sensitivity and specificity. Each item represents symptoms of depression and describes a participant's condition in the preceding week; the participants answer each item with either 'yes' or 'no'. All items are summed (total score 0-15). A score of six or greater is a cutoff for depression. The GDS has a Cronbach's alpha of 0.78.
Change in the participants' level of health-related quality of life | Change from baseline (T0) to immediately (T1), 6 months (T2) and 12 months (T3) after completion of the intervention
  Participants' health-related quality of life (HRQoL) will be measured by the Chinese version of the Stroke-Specific Quality of Life Scale (SSQOL-C), which has 47 items with 11 domains ranging from physical to psychosocial and participation. The items are about the health conditions of the participants and how much difficulty the participants have when doing everyday self-care tasks. The items are scored from 1 - 'strongly disagree/cannot do it' to 5 - 'strongly agree/no trouble'. Total score is yielded by summing all item scores (range 47-235): the higher the score, the higher the HRQoL. It has acceptable internal consistency (Cronbach's alpha: 0.63-0.93) and convergent validity.
Change in the participants' level of satisfaction with the performance of self-management behaviours | Change from baseline (T0) to immediately (T1), 6 months (T2) and 12 months (T3) after completion of the intervention
  The 11-item Chinese version of the Stroke Self-management Behaviours Performance Scale (SSBPS-C) will be adopted to assess participants' satisfaction with the performance of self-management behaviours. Each item is scored using a range from 0 - 'very dissatisfied' to 10 - 'very satisfied'. Taking the sum of all item scores yields one total score (range 0-110), and the higher the score, the higher the satisfaction. This scale has a Cronbach's alpha of 0.93.
Change in the participants' level of self-efficacy | Change from baseline (T0) to immediately (T1), 6 months (T2) and 12 months (T3) after completion of the intervention
  The Chinese version of the Stroke Self-Efficacy Questionnaire (SSEQ-C) will be used to measure self-efficacy. It has 13 items, each is scored using a scale from 0 - 'no confidence' to 10 - 'very confident'. The items are about the participants' perceived extent of confidence in doing everyday activities and self-management tasks. A total score is yielded by summing all items (range 0-130). A higher total score represents higher self-efficacy. The scale has acceptable internal consistency (Cronbach's alpha=0.92) and convergent validity.
Change in the participants' level of outcome expectation | Change from baseline (T0) to immediately (T1), 6 months (T2) and 12 months (T3) after completion of the intervention
  The Chinese version of the Stroke Self-management Outcome Expectation Scale (SSOES-C) will be used to measure the participants' outcome expectation beliefs. It has 11 items, each rated using a scale from 0 - 'strongly disagree' to 10 - 'strongly agree'. The score of each item indicates the participants' confidence in the expected outcomes to occur. All item scores will be calculated by summation (total score 0-110). A higher score represents higher outcome expectations. This scale has good internal consistency (Cronbach's alpha=0.94).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lo, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Suzanne Lo, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo SHS, Chau JPC, Choi KC, Shum EWC, Yeung JHM, Li SH. Promoting community reintegration using narratives and skills building for young adults with stroke: a protocol for a randomised controlled trial. BMC Neurol. 2021 Jan 4;21(1):3. doi: 10.1186/s12883-020-02015-5. PMID 33397316